CLINICAL TRIAL: NCT06487013
Title: A Pivotal Study to Evaluate the Effectiveness and Safety of ArcBlate Palliative Treatment for Patients With Painful Bone Metastases
Brief Title: Effectiveness and Safety of ArcBlate Palliative Treatment for Patients With Painful Bone Metastases: A Pivotal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: EpiSonica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTP-BM-22-01
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Bone Metastases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MRgHIFU treatment arm (Experimental): Subjects will be randomized to MRgHIFU treatment arm and will pass the Screening Fail criteria preceded in normal fashion to MRgHIFU treatment at the same session.
  Interventions: Device: ArcBlate Focused Ultrasound Ablation System
- Sham treatment arm (Sham Comparator): Subjects who will be randomized to sham treatment arm and passed the Screening Fail Criteria (i.e. MRI Screening and Sonication Screening) will undergo a sham MRgHIFU treatment with sonication energy disabled.
  Interventions: Other: Sham MRgHIFU treatment

INTERVENTIONS:
Device: ArcBlate Focused Ultrasound Ablation System — MR-guided High Intensity Focused Ultrasound (MRgHIFU)
  Arms: MRgHIFU treatment arm
Other: Sham MRgHIFU treatment — Sham MRgHIFU treatment
  Arms: Sham treatment arm

SUMMARY:
A Pivotal Study to Evaluate the Effectiveness and Safety of ArcBlate Palliative Treatment for Patients With Painful Bone Metastases

DETAILED DESCRIPTION:
Pain palliation of bone metastasis through localized denervation by thermal ablation.

ELIGIBILITY:
Inclusion Criteria:

* Provisional Screening (Screening 1):

  1. Men and women aged 18 and older.
  2. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at enrollment.
  3. Patients who are able and willing to give consent and able to attend all study visits.
  4. Patients who are suffering from painful bone metastases.
  5. Patients who refuse other accepted available treatments such as surgery or radiotherapy for pain palliation.
  6. Patient with NRS (0-10 scale) pain score ≥ 4 irrespective of medication.
  7. Able to communicate sensations during the ArcBlate MRgHIFU treatment.
  8. Patients on ongoing systemic anticancer treatment for at least 2 weeks before treatment:
* with same systemic anticancer treatment (as documented from patient medical dossier), And
* worst pain NRS still ≥ 4, And
* do NOT plan to initiate a new chemotherapy for pain palliation throughout the study duration.

  (9) No radiation therapy to targeted (most painful) lesion in the past two weeks before treatment.

  (10) Bisphosphonate intake should remain stable throughout the study duration. (11) Patients will have from 1 to 5 painful lesions and only the most painful lesion will be treated.

  (12) Patients with persistent distinguishable pain associated with 1 site to be treated (if patient has pain from additional sites, the pain from the additional sites must be evaluated as being less intense by at least 2 points on the NRS compared to the site to be treated).
* MRI Screening (Screening 2):

  1. Targeted tumor(s) are ArcBlate MRgHIFU accessible and are located in ribs, extremities (excluding joints), pelvis, shoulders and in the posterior aspects of the following spinal vertebra: Lumbar vertebra (L3 - L5), Sacral vertebra (S1 - S5).
  2. Patient whose targeted (treated) lesion is on bone and the interface between the bone and lesion is deeper than 10-mm from the skin.
  3. Targeted (treated) tumor clearly visible by non-contrast MRI, and ArcBlate MRgHIFU accessible.
* Sonication Screening (Screening 3):

  1. Subjects could tolerate planned test sonications per randomized treatment.

Exclusion Criteria:

* Provisional Screening (Screening 1):

  (1) Patients who either
* need surgical stabilization of the affected bony structure (>7 fracture risk score), Or
* targeted tumor is at an impending fracture site (>7 on fracture risk score), Or
* patients with surgical stabilization of tumor site with metallic hardware. (2) Targeted (treated) lesion is in the skull. (3) Patients on dialysis. (4) Patients with life expectancy < 3-Months. (5) Patients with an acute medical condition (e.g., pneumonia, sepsis) that is expected to hinder them from completing this study.

  (6) Patients with unstable cardiac status including:
* Unstable angina pectoris on medication,
* Patients with documented myocardial infarction within six months of protocol entry,
* Congestive heart failure requiring medication (other than diuretic),
* Patients on anti-arrhythmic drugs. (7) Severe hypertension (diastolic blood pressure > 100 mmHg on medication). (8) Patients with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations (unable to fit into ArcBlate MRgHIFU), etc.

  (9) Patients with an active infection or severe hematological, neurological, or other uncontrolled disease.

  (10) Known intolerance or allergies to the MRI contrast agent (e.g., Gadolinium or Magnevist) and Computed Tomography (CT) contrast agent including advanced kidney disease.

  (11) Severe cerebrovascular disease (multiple CerebroVascular Accident (CVA) or CVA within 6 months).

  (12) Individuals who are not able or willing to tolerate the required prolonged stationary position during treatment (approximately 2 hrs.).

  (13) Are participating or have participated in another clinical trial in the last 30 days.

  (14) Patients initiating a new chemotherapy regime, or radiation (for the targeted most painful lesion) within the last 2 weeks before treatment.

  (15) Patients unable to communicate with the investigator and staff. (16) Patients with persistent undistinguishable pain (pain source unidentifiable).

  (17) The targeted tumor is less than 2 points more painful compared to other painful lesions on the site specific NRS.

  (18) Patients with calcified treatment area. (19) Pregnant women.
* MRI Screening (Screening 2):

  1. Target (treated) lesion is less than 10-mm from nerve bundles, bowels or bladder.
  2. Extensive scarring in the energy path of the planned treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-12-08 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Pain response rate to therapy at 30 days after treatment | at 30 days after treatment
  Pain response rate is assessed by composite endpoint of change from baseline in worst Numerical Rating Scale (NRS) pain score (0-10 scale) and morphine equivalent daily dose (MEDD) intake.
  Patients with Complete response (CR) or Partial response (PR) are defined as responders to therapy.
  1. Complete response (CR): Pain score 0 without analgesic increase.
  2. Partial response (PR): Pain reduction of 2 or more without analgesic increase; or analgesic reduction of 25% without pain increase.
  The proportion of responders of the subjects who completed treatment is defined as the pain response rate of this study.

SECONDARY OUTCOMES:
Change from baseline in NRS pain score (0-10 scale) | at 1, 3, 7, 14, 30, 60 and 90 days after treatment
  The changes of NRS pain score between post-treatment and pre-treatment. The pain NRS is a single 11-point numeric scale (0-10 scale), with 0 representing one pain extreme (e.g., "no pain") and 10 representing the other pain extreme (e.g., "pain as bad as you can imagine" and "worst pain imaginable").
Change from baseline in MEDD intake | at 7, 14, 30, 60 and 90 days after treatment
  The changes of MEDD intake between post-treatment and pre-treatment.
Change from baseline in Brief Pain Inventory (BPI-QoL) | at 30, 60 and 90 days after treatment
  The changes of BPI between post-treatment and pre-treatment. The BPI is used to rapidly assess the severity of pain and the impact of pain on daily functions.
  The BPI has seven interference items, such as general activity, mood, walking ability, normal work (including housework), relations with other people, sleep, and enjoyment of life. The assessment areas of the BPI include severity of pain, impact of pain on daily function, location of pain, pain medications and amount of pain relief in the past 24 hours or the past week.
Pain response rate to therapy | at 60 and 90 days after treatment
  Patients with Complete response (CR) or Partial response (PR) are defined as responders to therapy.
Quality of Life as measured by EORTC QLQ-C15-PAL questionnaire | at 30, 60 and 90 days after treatment
  The QLQ-C15-PAL contains seven symptom scales (dyspnoea, pain, insomnia, fatigue, appetite loss, nausea and vomiting, and constipation) and three functional scales (physical functioning, emotional functioning, and overall QoL), which were identified as being relevant to the palliative population. Items on the QLQ-C15-PAL questionnaire are rated from 1 (not at all) to 4 (very much), with the exception of the overall QoL status item, which was rated from 1 (very poor) to 7 (excellent). A higher score for the symptom scales represents a higher level of symptomatology and, therefore, a decreased QoL. By contrast, a higher score for the functional scales represents a higher level of functionality and, therefore, an increased QoL. Each scale was transformed to a score ranging from 0 to 100, according to their respective scoring manual.
Total number of Adverse Events (AEs) | within the first 90 days within treatment
  Total numbers of complications and AEs, including unintended lesions that occur as a result of treatment with MR-HIFU.

CONTACTS AND LOCATIONS:
Locations (4):
- Taiwan (4):
  - Far Eastern Memorial Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital - Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No